CLINICAL TRIAL: NCT00195260
Title: Phase I Dose-Escalation Study Of Oral SKI-606 In Subjects With Advanced Malignant Solid Tumors
Brief Title: Study Evaluating SKI-606 (Bosutinib) In Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3160A1-100; B1871012
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-01

CONDITIONS: Neoplasms
Keywords: Solid tumors
MeSH Terms: conditions — Neoplasms | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose escalation (Experimental): Dose finding study of monotherapy bosutinib in patients with advanced solid tumors.
  Interventions: Drug: bosutinib
- Colorectal Cancer (Experimental): Enroll 30 patients at RP2D to further evaluate safety and efficacy in subgroup population.
  Interventions: Drug: bosutinib
- Pancreatic Cancer (Experimental): Enroll 30 patients at RP2D to further evaluate safety and efficacy in subgroup population.
  Interventions: Drug: bosutinib
- Non-Small Cell Lung Cancer (NSCLC) (Experimental): Enroll 30 patients at RP2D to further evaluate safety and efficacy in subgroup population.
  Interventions: Drug: bosutinib

INTERVENTIONS:
Drug: bosutinib — Dose levels evaluated 50mg, 100mg, 200mg, 300mg, 400mg, 500mg and 600mg. 500mg was identified as MTD, however due to GI toxicities at that dose, 400mg was selected as the RP2D. Drug was administered as long as tolerable and disease under study did not worsen.
  Arms: Dose escalation
Drug: bosutinib — 400mg QD bosutinib, as long as tolerated and disease under study does not worsen.
  Arms: Colorectal Cancer
Drug: bosutinib — 400mg QD bosutinib, as long as tolerated and disease under study does not worsen.
  Arms: Pancreatic Cancer
Drug: bosutinib — 400mg QD bosutinib, as long as tolerated and disease under study does not worsen.
  Arms: Non-Small Cell Lung Cancer (NSCLC)

SUMMARY:
To evaluate the safety and tolerability of oral SKI-606 (bosutinib) administered on a daily schedule to subjects with advanced malignant solid tumors and to define a maximum tolerated dose (MTD) in this subject population.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or recurrent solid malignancy confirmed histologically or cytologically for which no effective therapy is available.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
* Measurable disease as outlined by the modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Other inclusion applies.

Exclusion Criteria:

* Use of any systemic antitumor agents or any investigational agent within 28 days before the first dose of test article is administered.
* Prior exposure to SKI-606 or any other Src-kinase inhibitor, major surgery or radiotherapy within 14 days before the first dose of test article (recovery from previous surgery should be complete before day 1).
* Active central nervous system (CNS) metastases, as indicated by clinical symptoms, cerebral edema, requirement for corticosteroids and/or progressive growth (Treated CNS metastases must be stable for >= 2 weeks before day 1).
* Other exclusion applies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2004-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (16):
  - Pfizer Investigational Site, Birmington, Alabama
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Indianpolis, Indiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Lansing, Michigan
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, UNC Chapel Hill, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Tyler, Texas
  - Pfizer Investigational Site, Seattle, Washington

REFERENCES:
- [Derived] Hsyu PH, Mould DR, Abbas R, Amantea M. Population pharmacokinetic and pharmacodynamic analysis of bosutinib. Drug Metab Pharmacokinet. 2014;29(6):441-8. doi: 10.2133/dmpk.DMPK-13-RG-126. Epub 2014 Jun 10. PMID 24919837 (Retraction: PMID 30922682 Drug Metab Pharmacokinet. 2019 Apr;34(2):163)

RESULTS

PARTICIPANT FLOW:
Groups:
- Bosutinib 50 mg: Bosutinib 50 milligram (mg) capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
- Bosutinib 100 mg: Bosutinib 100 mg capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
- Bosutinib 200 mg: Bosutinib 200 mg capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
- Bosutinib 300 mg: Bosutinib 300 mg capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
- Bosutinib 400 mg: Bosutinib 400 mg capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
- Bosutinib 500 mg; Maximum Tolerated Dose (MTD) lead-in: Bosutinib 500 mg capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
- Bosutinib 600 mg: Bosutinib 600 mg capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
- Colorectal Cancer: Participants with colorectal cancer received bosutinib 400 mg capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
- Pancreatic Cancer: Participants with pancreatic cancer received bosutinib 400 mg capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
- Non-small Cell Lung Cancer (NSCLC): Participants with NSCLC received bosutinib 400 mg capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
Period: Part 1: Dose Escalation
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg | Maximum Tolerated Dose (MTD) lead-in | Colorectal Cancer | Pancreatic Cancer | Non-small Cell Lung Cancer (NSCLC)
Started | 4 | 4 | 6 | 7 | 7 | 7 | 10 | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 6 | 7 | 7 | 7 | 10 | 6 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Disease Progression | 3 | 2 | 5 | 6 | 4 | 6 | 7 | 4 | 0 | 0 | 0
Not completed — Symptomatic Deterioration | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Recommended Phase 2 Dose (RP2D)
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg | Maximum Tolerated Dose (MTD) lead-in | Colorectal Cancer | Pancreatic Cancer | Non-small Cell Lung Cancer (NSCLC)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 37 | 38 | 25
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 38 | 23
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 29 | 15
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Participants received bosutinib capsule orally once daily continuously in 21-day cycles in dose escalation schemes of 50 mg, 100 mg, 200 mg, 300 mg, 400 mg, 500 mg, 600 mg, MTD-lead in (500 mg) until disease progression, unacceptable toxicity, or consent withdrawal.
- RP2D 400 mg: Participants with colorectal cancer, pancreatic cancer, NSCLC received RP2D of bosutinib (400 mg) capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
- Total: Total of all reporting groups
Arm/Group | Part 1 | RP2D 400 mg | Total
Number analyzed (Participants) | 51 | 100 | 151
Age Continuous [Mean (Standard Deviation); unit: years] | 57.00 (12.67) | 60.30 (11.48) | 59.10 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 (participants) | 54 | 83
  Male | 22 | 46 | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT) in Part 1
Description: DLT included any grade 3 or 4 clinically-evident non-hematologic toxicity, grade 4 neutropenia of greater than or equal to (>=) 7-day duration or with fever >= 38.5 degrees Celsius (febrile neutropenia); grade 4 thrombocytopenia >= 2-day duration or with bleeding requiring platelet transfusion, any clinically-significant grade >= 2 toxicity that requires >=14 days to resolve (to less than or equal to [=<] grade 1) which occurred in first 21 days of study and considered at least possibly related to bosutinib.
Time Frame: Part 1 Baseline up to Day 28
Population: Safety population included all participants enrolled in a dose escalation cohort who had taken at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- MTD-lead in: Bosutinib 500 mg capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg | MTD-lead in
Number analyzed (Participants) | 4 | 4 | 6 | 7 | 7 | 7 | 10 | 6
participants | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0

2. Primary Outcome: Number of Participants With Adverse Events (AEs) by Seriousness
Description: Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: Baseline up to 30 days after last dose
Population: Safety population included all participants who had taken at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg | MTD-lead in | RP2D 400 mg
Number analyzed (Participants) | 4 | 4 | 6 | 7 | 7 | 7 | 10 | 6 | 100
participants
  AEs | 4 | 4 | 6 | 7 | 7 | 7 | 10 | 6 | 100
  Serious adverse events (SAEs) | 4 | 3 | 2 | 3 | 5 | 2 | 7 | 3 | 47

3. Primary Outcome: Duration of Most Frequently Observed Adverse Events (AEs)
Description: The most frequently observed treatment-emergent AEs were gastrointestinal disorders which included diarrhea, nausea and vomiting. Duration of AE per event is calculated as AE stop date minus AE start date plus 1.
Time Frame: Baseline up to 30 days after last dose
Population: Safety population included all participants who had taken at least 1 dose of study medication.
Measure: Median (Full Range); unit: days
Groups:
- MTD lead-in: Bosutinib 500 mg capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg | MTD lead-in | RP2D 400 mg
Number analyzed (Participants) | 4 | 4 | 6 | 7 | 7 | 7 | 10 | 6 | 100
days
  Diarrhea | 1.0 [1 to 1] | NA [NA to NA] — Data was not analyzed as no participants reported the event in this particular cohort. | 12.0 [1 to 27] | 2.0 [1 to 15] | 3.5 [1 to 7] | 7.0 [1 to 33] | 1.0 [1 to 23] | 1.0 [1 to 30] | 3.0 [1 to 75]
  Nausea | 2.0 [1 to 14] | 1.0 [1 to 11] | 1.0 [1 to 8] | 9.0 [1 to 366] | 4.0 [1 to 15] | 7.0 [1 to 94] | 3.0 [1 to 24] | 7.0 [1 to 24] | 13.0 [1 to 126]
  Vomiting | 2.5 [1 to 4] | 1.0 [1 to 9] | NA [NA to NA] — Data was not analyzed as no participants reported the event in this particular cohort. | 1.0 [1 to 13] | 3.0 [1 to 5] | 1.0 [1 to 3] | 2.0 [1 to 24] | 2.5 [1 to 9] | 2.0 [1 to 62]

4. Primary Outcome: Number of Participants With Best Overall Response (BOR) in Part 1
Description: BOR:investigator assessment by modified Response Evaluation Criteria in Solid Tumors (RECIST), recorded from treatment start until disease progression/recurrence. Complete Response:disappearance of all lesions. Partial Response (PR):>=30% decrease in sum of longest diameters (SLDs) of target lesions (TLs) taking as reference baseline SLD. Progressive disease (PD):>=20% increase in SLD of TLs taking as reference smallest SLD since treatment start, or appearance of >=1 new lesion. Stable disease: neither shrinkage for PR nor increase for PD taking as reference smallest SLD since treatment start.
Time Frame: Part 1 Baseline, last week (Day 15 to 23) of cycles 2, 4, 6, 8 and thereafter every 3 cycles up to 30 days after last dose
Population: Efficacy evaluable population: participants who received at least 1 cycle (15 doses) of study medication, had no eligibility violations, did not use prohibited anti-cancer treatment, had baseline disease assessment, at least 1 disease assessment post-baseline/had experienced clinical progression/death before first post-baseline disease assessment.
Measure: Number; unit: participants
Groups:
- Bosutinib 500 mg: Bosutinib 600 mg capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
- Bosutinib 600 mg; MTD-lead in: Bosutinib 500 mg capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg | MTD-lead in
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 6 | 4 | 3
participants
  Complete response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial response | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Stable disease | 0 | 2 | 2 | 5 | 3 | 2 | 4 | 2
  Progressive disease | 3 | 1 | 4 | 1 | 2 | 3 | 0 | 1
  Indeterminate | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Not done | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Best Overall Response (BOR) in Part 2
Description: BOR: investigator assessment by modified RECIST, recorded from treatment start until disease progression/recurrence. Complete Response: disappearance of all lesions. PR: >=30% decrease in SLDs of TLs taking as reference baseline SLD. PD: >=20% increase in SLD of TLs taking as reference smallest SLD since treatment start, or appearance of >=1 new lesion. Stable disease: neither shrinkage for PR nor increase for PD taking as reference smallest SLD since treatment start.
Time Frame: Part 2 Baseline, last week (Day 15 to 23) of cycles 2, 4, 6, 8 and thereafter every 3 cycles up to 30 days after last dose
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Colorectal Cancer | Pancreatic Cancer | Non-small Cell Lung Cancer (NSCLC)
Number analyzed (Participants) | 34 | 22 | 19
participants
  Complete response | 0 | 0 | 0
  Partial response | 0 | 0 | 0
  Stable disease | 10 | 3 | 9
  Progressive disease | 24 | 18 | 9
  Indeterminate | 0 | 0 | 0
  Not done | 0 | 1 | 1

6. Primary Outcome: Maximum Tolerated Dose (MTD) in Part 1
Description: MTD: highest dose level at which not more than 1 of 6 participants experienced DLT after 21 days of treatment (Cycle 1). DLT included any grade 3 or 4 clinically-evident non-hematologic toxicity, grade 4 neutropenia of >= 7-day duration or with fever >= 38.5 degrees Celsius (febrile neutropenia); grade 4 thrombocytopenia >= 2-day duration or with bleeding requiring platelet transfusion, any clinically-significant grade >= 2 toxicity that requires >=14 days to resolve (to =< grade 1) which occurred in first 21 days of study and considered at least possibly related to bosutinib.
Time Frame: Part 1 Day 1 up to Day 28
Population: as for outcome 1
Measure: Number; unit: mg
Groups:
- All Participant: All participants who received bosutinib capsule (50 mg, 100 mg, 200 mg, 300 mg, 400 mg, 500 mg, 600 mg, MTD-lead in) orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal.
Arm/Group | All Participant
Number analyzed (Participants) | 51
mg | 500

7. Secondary Outcome: Maximum Tolerated Dose (MTD) for Prolonged Use
Description: MTD for prolonged use was the highest dose level at which not more than 1 of 6 participants experienced DLT after 21 days of treatment (Cycle 1) and was selected as recommended dose in Phase 2, due to substantial number of Grade 2 gastrointestinal toxicities observed in the MTD lead-in cohort (500 mg).
Time Frame: Part 1 Day 1 up to Day 28
Population: as for outcome 1
Measure: Number; unit: mg
Arm/Group | All Participant
Number analyzed (Participants) | 51
mg | 400

8. Secondary Outcome: Number of Participants With Change From Baseline in Laboratory Test Results
Description: Criteria for potentially clinically significant (PCS) laboratory values: albumin <20, hemoglobin <80 gram/liter(g/L); alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase >5*upper limit of normal(ULN) milliunit/milliliter(mU/mL); bilirubin total, creatinine>3*ULN micromole/L; calcium <1.75 and >3.1,potassium <3 and >6, sodium <130, glucose <2.2,phosphorous <0.6 millimole/L; international normalized ratio >2*ULN, partial thromboplastin time, prothrombin time >2*ULN seconds; platelet count <50*10^9/L. Participants meeting at least 1 PCS criteria are reported.
Time Frame: Baseline up to end of treatment (Week 95)
Population: Safety population included all participants who had taken at least 1 dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable (at least 1 on-therapy laboratory assessment) for this measure for each group respectively.
Measure: Number; unit: participants
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg | MTD-lead in | RP2D 400 mg
Number analyzed (Participants) | 4 | 4 | 6 | 7 | 7 | 7 | 8 | 6 | 96
participants
  Albumin (<20 g/L) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Alkaline phosphatase (>5*ULN) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 5
  Bilirubin total (>3*ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Calcium (<1.75 mmol/L) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Calcium (>3.1 mmol/L) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine (>3*ULN) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Glucose (<2.2 mmol/L) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Phosphorus (<0.6 mmol/L) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Potassium (<3 mmol/L) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Potassium (>6 mmol/L) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Aspartate aminotransferase (> 5*ULN)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5
  Alanine aminotransferase (> 5*ULN) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5
  Sodium (<130 mmol/L) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 7
  International normalized ratio (>2*ULN) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 6
  Prothrombin time (>2*ULN) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 7
  Partial thromboplastin time (>2*ULN) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1
  Hemoglobin (<80 g/L) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Platelets (<50*10^9/L) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0

9. Secondary Outcome: Number of Participants With Change From Baseline in Electrocardiogram (ECG) and Chest X-ray
Description: Number of participants with PCS ECG findings is reported on-therapy (OT) and at final visit (FV). Criteria for PCS ECG findings: heart rate (HR) =<45 beats/minute (bpm) and decrease (Dec) >15/>=120 bpm and decrease of >15 bpm; PR interval (Int) >=220 millisecond (msec), increase (Inc) >=20 msec, QRS Int >=120 msec, corrected QT (QTc) and QTc using fridericia formula(QTcF) Int >500 msec, increase >60 msec; no sinus rhythm; overall ECG abnormal. Participants with at least 1 measurement exceeding the criteria for PCS are reported.
Time Frame: Baseline up to end of treatment (Week 95)
Population: Safety population included all participants who had taken at least 1 dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable (at least 1 on-therapy assessment) for this measure and 'n' represents participants evaluable under each category for each group respectively.
Measure: Number; unit: participants
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg | MTD-lead in | RP2D 400 mg
Number analyzed (Participants) | 4 | 4 | 6 | 7 | 7 | 7 | 10 | 6 | 93
participants
  OT: HR (<=45/Dec >15bpm) (n=4,4,6,7,7,7,10,6,93) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  OT: HR (>=120/Inc >15bpm) (n=4,4,6,7,7,7,10,6,93) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  OT:PR Int(>=220/Inc>20msec)(n=4,4,6,7,7,7,10,6,93) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  OT: QRS Int (>=120 msec) (n=4,4,6,7,7,7,10,6,93) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 8
  OT: QTc Int (Inc >60 msec) (n=4,4,6,7,7,7,10,6,93) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  OT: QTc Int (>500 msec) (n=4,4,6,7,7,7,10,6,93) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  OT: QTcF Int (Inc >60 msec) (n=0,0,0,0,0,0,1,3,89) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  OT: QTcF Int (>500 msec) (n=0,0,0,0,0,0,1,3,89) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  OT: No sinus rhythm (n=4,4,6,7,7,7,10,6,93) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29
  OT: Overall ECG abnormal (n=4,4,6,7,7,7,10,6,93) | 3 | 4 | 5 | 7 | 6 | 6 | 8 | 6 | 63
  FV: HR (>=120/Inc >15bpm) (n=1,2,2,4,3,4,3,1,42) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  FV:PR Int(>=220/Inc >20msec)(n=1,2,3,4,3,4,3,1,42) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  FV: QRS Int (>=120 msec) (n=1,2,2,4,3,4,3,1,42) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4
  FV: QTc Int (>500 msec) (n=1,2,3,4,3,4,3,1,42) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  FV: No sinus rhythm (n=1,2,2,4,3,4,3,1,42) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  FV: Overall ECG abnormal (n=1,2,3,4,3,4,3,1,42) | 1 | 1 | 1 | 0 | 2 | 3 | 3 | 1 | 18
  Chest X-ray (n=0,0,0,0,0,0,0,0,0) | NA — Data for this pre-specified category was collected but not statistically summarized for analysis as there were no clinically significant changes observed. | NA — Data for this pre-specified category was collected but not statistically summarized for analysis as there were no clinically significant changes observed. | NA — Data for this pre-specified category was collected but not statistically summarized for analysis as there were no clinically significant changes observed. | NA — Data for this pre-specified category was collected but not statistically summarized for analysis as there were no clinically significant changes observed. | NA — Data for this pre-specified category was collected but not statistically summarized for analysis as there were no clinically significant changes observed. | NA — Data for this pre-specified category was collected but not statistically summarized for analysis as there were no clinically significant changes observed. | NA — Data for this pre-specified category was collected but not statistically summarized for analysis as there were no clinically significant changes observed. | NA — Data for this pre-specified category was collected but not statistically summarized for analysis as there were no clinically significant changes observed. | NA — Data for this pre-specified category was collected but not statistically summarized for analysis as there were no clinically significant changes observed.

10. Secondary Outcome: Concomitant Medications Used for Management of Adverse Events (AEs)
Description: Number of participants taking any non-study medications which were administered from Day 1 up to end of treatment (Week 95) as a management of an AE was to be reported.
Time Frame: Day 1 up to end of treatment (Week 95)
Population: Data for this pre-specified outcome measure was not statistically summarized for analysis, but collected and reported in individual participant listings as planned.
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg | MTD-lead in | RP2D 400 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Karnofsky Performance Score
Description: Karnofsky performance score is used to quantify participant's general well-being and activities of daily life and participants are classified based on their functional impairment. Karnofsky performance score is 11 level score which ranges between 0 (death) to 100 (complete healthy status). Higher score means higher ability to perform daily tasks.
Time Frame: Baseline up to end of treatment (Week 95)
Population: Data for this pre-specified outcome was collected but not statistically summarized for analysis as there were no clinically significant changes observed.
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg | MTD-lead in | RP2D 400 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Change From Baseline in Physical Examination
Description: Physical examinations included body weight, height and vital signs and only finding that exceeded the criterion for PCS was weight. Criteria for weight was: an increase or decrease of >=10% from baseline.
Time Frame: Baseline up to end of treatment (Week 95)
Population: Safety population included all participants who had taken at least 1 dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable (at least 1 on-therapy assessment) for this measure for each group respectively.
Measure: Number; unit: participants
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg | MTD-lead in | RP2D 400 mg
Number analyzed (Participants) | 4 | 4 | 6 | 7 | 7 | 7 | 7 | 6 | 87
participants
  Weight (decrease >=10%) | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 3
  Weight (increase >=10%) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 3

13. Secondary Outcome: Number of Participants With Change From Baseline in Opthalmologic Examination
Description: Ophthalmologic evaluation included visual acuity, funduscopic examination, and any clinically-significant abnormality.
Time Frame: Baseline up to end of treatment (Week 95)
Population: Safety population included all participants who had taken at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg | MTD-lead in | RP2D 400 mg
Number analyzed (Participants) | 4 | 4 | 6 | 7 | 7 | 7 | 10 | 6 | 100
participants | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4

14. Secondary Outcome: Overall Survival (OS) in Part 2
Description: Time in weeks from the start of study treatment to date of death due to any cause. OS was calculated as (the death date minus the date of first dose of study medication plus 1) divided by 7. Death was determined from death case report forms (CRFs) or from follow-up contact data (where the participant current status was death).
Time Frame: Part 2 Baseline until death or 3, 6, 9 and 12 months after treatment discontinuation
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Colorectal Cancer | Pancreatic Cancer | Non-small Cell Lung Cancer (NSCLC)
Number analyzed (Participants) | 34 | 22 | 19
weeks | 27.7 [23.0 to 34.3] | 14.7 [8.1 to 22.9] | 34.0 [16.7 to 55.0]

15. Secondary Outcome: Progression Free Survival (PFS) in Part 2
Description: Time in weeks from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for PD, or from death CRFs).
Time Frame: Part 2 Baseline until death or 3, 6, 9 and 12 months after treatment discontinuation
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Colorectal Cancer | Pancreatic Cancer | Non-small Cell Lung Cancer (NSCLC)
Number analyzed (Participants) | 34 | 22 | 19
weeks | 6.0 [5.3 to 7.1] | 6.0 [5.3 to 6.1] | 5.7 [5.3 to 19.3]

16. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 hour (pre-dose) on Day 1, 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24 (0 hour [pre-dose] on Day 15) hours post-dose on Day 14
Population: Analysis population included all participants who had taken at least 1 dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants evaluable for specific time points.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Groups:
- Bosutinib 400 mg (Part 1 + Part 2): Bosutinib 400 mg capsule orally once daily continuously in 21-day cycles until disease progression, unacceptable toxicity, or consent withdrawal in both Part 1 and Part 2 participants.
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg (Part 1 + Part 2) | Bosutinib 500 mg | Bosutinib 600 mg
Number analyzed (Participants) | 4 | 4 | 6 | 7 | 69 | 13 | 10
nanogram/milliliter (ng/mL)
  Day 1 (n = 4, 4, 6, 7, 54, 13, 10) | 4.89 (3.69) | 17.0 (9.75) | 43.1 (26.9) | 63.7 (34.7) | 117.0 (69.0) | 125.0 (63.2) | 206.0 (190.0)
  Day 15 (n = 3, 4, 5, 5, 69, 10, 2) | 6.92 (3.07) | 19.6 (3.31) | 95.4 (60.0) | 76.6 (37.0) | 190.0 (116.0) | 273.0 (197.0) | 304.0 (NA) — Standard deviation obtained by sampling distribution of 2 participants was not meaningful, hence not reported.

17. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 hour (pre-dose) on Day 1, 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24 (0 hour [pre-dose] on Day 15) hours post-dose on Day 14
Population: Analysis population included all participants who had taken at least one dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants evaluable for specific time points.
Measure: Median (Full Range); unit: hours
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg (Part 1 + Part 2) | Bosutinib 500 mg | Bosutinib 600 mg
Number analyzed (Participants) | 4 | 4 | 6 | 7 | 69 | 13 | 10
hours
  Day 1 (n = 4, 4, 6, 7, 54, 13, 10) | 6.01 [4.00 to 8.00] | 4.08 [2.00 to 6.00] | 6.00 [2.05 to 8.00] | 6.00 [3.23 to 6.17] | 4.00 [1.00 to 8.68] | 4.00 [2.00 to 8.00] | 6.00 [1.30 to 8.00]
  Day 15 (n = 3, 4, 5, 5, 69, 10, 2) | 4.00 [3.00 to 6.00] | 3.50 [2.25 to 4.03] | 4.00 [3.00 to 6.10] | 4.02 [3.00 to 6.00] | 4.00 [1.00 to 8.33] | 5.00 [1.00 to 8.00] | 3.53 [3.00 to 4.05]

18. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 hour (pre-dose) on Day 1, 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24 (0 hour [pre-dose] on Day 15) hours post-dose on Day 14
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg (Part 1 + Part 2) | Bosutinib 500 mg | Bosutinib 600 mg
Number analyzed (Participants) | 4 | 4 | 6 | 7 | 69 | 13 | 10
hours
  Day 1 (n = 3, 4, 6, 7, 47, 13, 10) | 12.86 (7.36) | 18.61 (4.91) | 20.80 (6.07) | 17.12 (6.01) | 18.63 (7.67) | 21.87 (7.39) | 19.94 (5.47)
  Day 15 (n = 3, 4, 5, 4, 53, 9, 2) | 25.84 (12.26) | 64.65 (67.31) | 30.04 (20.13) | 19.35 (7.54) | 19.89 (16.72) | 23.25 (15.00) | 16.29 (NA) — Standard deviation obtained by sampling distribution of 2 participants was not meaningful, hence not reported.

19. Secondary Outcome: Area Under the Concentration-Time Curve (AUC)
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption. Steady state concentration was achieved at Day 15.
Time Frame: 0 hour (pre-dose) on Day 1, 0 (pre-dose), 1, 2, 3, 4, 6, 8, 24 (0 hour [pre-dose] on Day 15) hours post-dose on Day 14
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg (Part 1 + Part 2) | Bosutinib 500 mg | Bosutinib 600 mg
Number analyzed (Participants) | 4 | 4 | 6 | 7 | 69 | 13 | 10
ng*hour/mL
  Day 1 (n = 3, 4, 6, 7, 47, 13, 10) | 129.0 (131.0) | 284.0 (72.8) | 920.0 (338.0) | 1200.0 (736.0) | 2340.0 (1230.0) | 2950.0 (1470.0) | 4300.0 (3310.0)
  Day 15 (n = 3, 4, 5, 4, 58, 9, 2) | 114.0 (33.3) | 329.0 (58.1) | 1670.0 (1130.0) | 1170.0 (699.0) | 2900.0 (1700.0) | 3580.0 (1820.0) | 4220.0 (NA) — Standard deviation obtained by sampling distribution of 2 participants was not meaningful, hence not reported.

20. Other Pre Specified Outcome: Gene Expression at Baseline
Description: Gene expression profile was evaluated by measuring transcript levels of messenger RNA (mRNA) in peripheral blood samples. Expression profiling of mRNA: done to measure the expressed genome of mRNA transcripts or done in a gene-specific targeted manner.
Time Frame: Baseline
Population: Data was not analyzed as the analysis was cancelled due to lack of samples provided from sites.
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg | MTD-lead in
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Bosutinib 50 mg | Bosutinib 100 mg | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg | MTD lead-in | RP2D 400 mg
Serious Adverse Events (participants affected / at risk) | 4/4 | 3/4 | 2/6 | 3/7 | 5/7 | 2/7 | 7/10 | 3/6 | 47/100
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 6/6 | 7/7 | 7/7 | 7/7 | 10/10 | 6/6 | 99/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib 50 mg (N=4) | Bosutinib 100 mg (N=4) | Bosutinib 200 mg (N=6) | Bosutinib 300 mg (N=7) | Bosutinib 400 mg (N=7) | Bosutinib 500 mg (N=7) | Bosutinib 600 mg (N=10) | MTD lead-in (N=6) | RP2D 400 mg (N=100)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Systemic candida (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib 50 mg (N=4) | Bosutinib 100 mg (N=4) | Bosutinib 200 mg (N=6) | Bosutinib 300 mg (N=7) | Bosutinib 400 mg (N=7) | Bosutinib 500 mg (N=7) | Bosutinib 600 mg (N=10) | MTD lead-in (N=6) | RP2D 400 mg (N=100)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 3 | 3 | 1 | 2 | 1 | 20
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 0 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 3
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Orbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0 | 2 | 4 | 3 | 9 | 3 | 51
Nausea (Gastrointestinal disorders) | 3 | 3 | 3 | 4 | 5 | 6 | 8 | 4 | 65
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 4 | 4 | 5 | 5 | 7 | 4 | 48
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 1 | 3 | 3 | 1 | 12
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 3 | 1 | 5 | 1 | 27
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 3 | 2 | 2 | 3 | 15
Eructation (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 1 | 3 | 2 | 1 | 15
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 12
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 7
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gastrointestinal oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 4 | 4 | 5 | 4 | 8 | 5 | 47
Oedema peripheral (General disorders) | 2 | 1 | 3 | 0 | 3 | 2 | 2 | 1 | 14
Pyrexia (General disorders) | 2 | 1 | 0 | 1 | 3 | 0 | 3 | 2 | 13
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 5
Early satiety (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2
Catheter thrombosis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 6
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 6
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Crepitations (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Nodule (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 4
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6
Temperature intolerance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 10
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
Viral pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 5
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 2 | 3 | 3 | 1 | 1 | 0 | 16
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 1 | 0 | 2 | 2 | 0 | 16
Breath sounds abnormal (Investigations) | 0 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 0 | 14
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 14
Pulmonary function test decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 12
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 10
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood urea decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 2 | 4 | 1 | 5 | 5 | 43
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 1 | 1 | 0 | 3 | 1 | 6
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 21
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 8
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 6
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 2 | 2 | 0 | 4 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 2 | 2 | 1 | 2 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 8
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cervix neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 2 | 4 | 0 | 2 | 3 | 2 | 11
Headache (Nervous system disorders) | 1 | 0 | 2 | 2 | 3 | 1 | 5 | 1 | 16
Cervical cord compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 5
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 1 | 1 | 6 | 2 | 2 | 11
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 4 | 2 | 3
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 4
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 4
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 2
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anger (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 3 | 0 | 3 | 2 | 23
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 22
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.